CLINICAL TRIAL: NCT01575665
Title: CO2 Rebreathing by a Partial Rebreathing Mask as a Treatment of Chronic Idiopathic Hyperventilation - a Pilot Study
Brief Title: Normalizing CO2 in Chronic Hyperventilation by a Novel Breathing Mask: A Pilot Study
Acronym: HVMASKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Rehaler (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8313-86
Record Dates: First submitted 2012-04-10; First posted 2012-04-11 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Hyperventilation; Chronic Idiopathic Hyperventilation; Dysfunctional Breathing; Respiratory Alkalosis
Keywords: Hyperventilation; Chronic Idiopathic Hyperventilation; Dysfunctional Breathing; Respiratory Alkalosis; Respiratory Acidosis
MeSH Terms: conditions — Hyperventilation; Alkalosis, Respiratory; Acidosis, Respiratory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Partial Rebreathing Mask (Experimental): A novel membrane breathing mask which facilitates a partial rebreathing of expired gas (thereby raising systemic CO2), while allowing a diffusion of oxygen from the atmosphere to the user, through the membranes.
  Interventions: Device: Partial Rebreathing Mask

INTERVENTIONS:
Device: Partial Rebreathing Mask — Inducing normal CO2 for two hours a day for four weeks
  Other Names: CDA mask; Balancair Mask

SUMMARY:
Background: Chronic Idiopathic Hyperventilation (CIH) is a form of dysfunctional breathing which has proven hard to treat effectively. The investigators hypothesised that by periodically inducing normocapnia over several weeks, it would be possible to raise the normal resting level/set point of CO2 and achieve a reduction of symptoms.

Methods: Six CIH patients were treated two hours a day for four weeks with a novel breathing mask. The mask was used to induce normocapnia in these chronically hypocapnic patients.

Capillary blood gases (PcCO2, pH, Standard Base Excess (SBE) etc.) were measured at baseline and once each week at least three hours after mask use, as well as spirometric values, breath holding tolerance and hyperventilation symptoms as per the Nijmegen Questionnaire (NQ),.

ELIGIBILITY:
Inclusion Criteria:

Chronic idiopathic hyperventilation, i.e.:

* PCO2 level below 4.7 kPa AND
* SBE value more negative than -1.0

Exclusion Criteria:

* Oxygen saturation of 95% or lower at rest

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Blood gas and acid/base status | Once every week in the treatment period of four weeks
  pH, PCO2, PO2, Standard Base Excess

SECONDARY OUTCOMES:
Hyperventilation symptoms | once a week
  Nijmegen Questionnaire
Breath Hold Tolerance | once a week
Spirometric values | once a week
  FEV1, FVC

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Dahl, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark